CLINICAL TRIAL: NCT06140628
Title: Clinical Study on 28 Day Continuous Improvement of Post-rejuvenation-treatment Skin With Formulations of A Proprietary Anti-aging Complex Composition
Brief Title: A 28-day Clinical Study on Facial Skin Rejuvenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Botanee Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: W23021025
Record Dates: First submitted 2023-10-31; First posted 2023-11-20 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Wrinkle; Skin Laxity; Skin Manifestations; Skin
MeSH Terms: conditions — Cutis Laxa; Skin Manifestations

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Formulation containing MLYAAT-1002® Composition (Active Comparator): After the Fotana4D Pro® treatment, daily use of the formulation for 28 days: apply one pump of the formulation to the treated side of the face in the morning and evening, respectively.
  Interventions: Combination Product: Fotona4D Pro® treatment followed by daily use of formulations containing MLYAAT-1002®
- Blank formulation without MLYAAT-1002® Composition (Placebo Comparator): After the Fotana4D Pro® treatment, daily use of the blank formulation for 28 days: apply one pump of the blank formulation to the control side of the face in the morning and evening, respectively.
  Interventions: Combination Product: Fotona4D Pro® treatment followed by daily use of formulations without MLYAAT-1002®

INTERVENTIONS:
Combination Product: Fotona4D Pro® treatment followed by daily use of formulations containing MLYAAT-1002® — Each subject will receive a single treatment of the Fotona4D Pro® , followed by the first application of the active comparator on the randomly assigned side of split-face (the treatment side) on the same day, and sequently, will apply the active comparator to this side twice a day for 28 days.
  Arms: Formulation containing MLYAAT-1002® Composition
Combination Product: Fotona4D Pro® treatment followed by daily use of formulations without MLYAAT-1002® — Each subject will receive a single treatment of the Fotona4D Pro® , followed by the first application of the placebo comparator on the randomly assigned side of split-face (the control side) on the same day, and sequently, will apply the placebo comparator to this side twice a day for 28 dayd.
  Arms: Blank formulation without MLYAAT-1002® Composition

SUMMARY:
This clinical trial aims to learn about the efficacy of MLYAAT-1002® (a proprietary anti-aging complex, MLYAAT is short for "multi-layer anti-ageing technology" ) in female subjects who have newly received the rejuvenation treatment by comparing visual clinical scores, skin attributes measurement and image analysis.

DETAILED DESCRIPTION:
The main expectation it aims to answer are:

* After the 4-week continuous use of the test skin product with MLYAAT-1002®, the skin aging problem is significantly improved compared with it of controlled product.
* After the single use of the test skin product with MLYAAT-1002®, the instant skin irritation after the Fotona4D Pro® treatment ( a nonablative fractional laser treatment for facial skin rejuvenation) is significantly lower compared with it of controlled product.
* After the 4-week continuous use of the test skin product with MLYAAT-1002®, the skin TEWL (transepidermal water loss) is significantly recovered from the Fotona4D Pro® treatment compared with it of controlled product. And the skin TEWL after the 4-week continuous use of test product is improved or not significantly worse than it before the Fotona4D Pro® treatment.
* After the 4-week continuous use of the test skin product with MLYAAT-1002®, no skin irritation symptom is worsen compared to it after the Fotona4D Pro® treatment.

ELIGIBILITY:
Inclusion Criteria:

* females aged 30-50
* no history of cosmetic allergies
* according to SKIN AGING ATLAS 2(Asian Type), the scores of under-eye wrinkles, pore appearance, forehead wrinkles are all > 2
* non-sensitive skin
* acceptable for split-face use of products for 28 days
* no using history of antibiotic in the past three months
* written informed consent and portrait right consent were obtained from all participants before study entry

Exclusion Criteria:

* subjects with known allergies or sensitivities to the ingredients in any of the study products
* anyone who is pregnant, nursing an infant, or planning a pregnancy during the study
* any symptoms of facial flushing, erythema, papules, desquamation, or edema as evaluated by a physician prior to initial screening or Fotona4D Pro treatment
* unhealed skin lesions
* participated in any other clinical trial within one month
* received facial skin treatments including but not limited to lasers, chemical peels, dermal fillers within one year
* taken/injected anti-allergy medication in the past one month
* other medical reasons that could affect the test results
* participants in other clinical trials at the same time

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2023-09-24 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2024-04-08 (Actual)

PRIMARY OUTCOMES:
changes in individual typology angle (ITA°) of facial skin | Day 0, Day 3, Day 7, Day 14, Day 28
  capturing facial images by VISIA-7 (CANFIELD, America) and calculating the ITA
changes in elasticity of facial skin (R2) | Day 0, Day 3, Day 7, Day 14, Day 28
  measuring gross elasticity (R2) by Cutometer® MPA580 (Courage&Khazaka, Germany)
changes in elasticity of facial skin (F4) | Day 0, Day 3, Day 7, Day 14, Day 28
  measuring firmness (F4) by Cutometer® MPA580 (Courage&Khazaka, Germany)
changes in facial skin topography (SEsm) | Day 0, Day 3, Day 7, Day 14, Day 28
  evaluating skin smoothness (SEsm) using VisioScan VC20（Courage&Khazaka，Germany）
changes in facial skin topography (SEw) | Day 0, Day 3, Day 7, Day 14, Day 28
  evaluating wrinkles (SEw) using VisioScan VC20（Courage&Khazaka，Germany）
changes in fine line depth of facial skin | Day 0, Day 3, Day 7, Day 14, Day 28
  evaluating peri orbital fine lines by Primos（CANFIELD, America）
changes in wrinkle depth of facial skin | Day 0, Day 3, Day 7, Day 14, Day 28
  evaluating crow's feet wrinkles by Primos（CANFIELD, America）
changes in skin thickness of facial skin | Day 0, Day 3, Day 7, Day 14, Day 28
  measuring skin thickness in µm by Ultrascan UC22（Courage&Khazaka，Germany）
changes in skin density of facial skin | Day 0, Day 3, Day 7, Day 14, Day 28
  measuring skin density (ultrasound density in % ) by Ultrascan UC22（Courage&Khazaka，Germany）

SECONDARY OUTCOMES:
changes in transepidermal water loss (TEWL，in g/m2/h) of facial skin | Day 0, Day 3, Day 7, Day 14, Day 28
  measuring the loss of water that passes from inside a body through the epidermis to the surrounding atmosphere by Tewameter® MPA580 (Courage&Khazaka，Germany)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoke Xu, Dr, Principal Investigator — Shenzhen Xiaoke BeauCare Clinic
Locations (1):
- Shanghai China-norm Quality Technical Service Co., Ltd., Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhang X, Ning M, Lin M, Tang Q, Liang Y, Wang F, Xu X. Continuous Skin Rejuvenation by Combining Nonablative Fractional Laser With Daily Application of a Multibeneficial Composition Formulation: A Blinded Randomized Clinical Trial Study. Health Sci Rep. 2025 Mar 2;8(3):e70423. doi: 10.1002/hsr2.70423. eCollection 2025 Mar. PMID 40041776